CLINICAL TRIAL: NCT02935036
Title: A Multi-center, Double-blind, Randomized, Placebo Controlled, Parallel-group Study to Evaluate the Efficacy and Safety of ADPS in the Treatment of Acne Vulgaris
Brief Title: Efficacy Study in Patients With Acne Vulgaris.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADPS 1602
Record Dates: First submitted 2016-10-12; First posted 2016-10-17 (Estimated); Results first posted 2018-09-18 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-09

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ADPS topical product (Experimental): A thin layer of study medication will be applied to cover affected areas once daily for 12 weeks
  Interventions: Drug: ADPS topical product
- Placebo Control (Placebo Comparator): A thin layer of study medication will be applied to cover affected areas once daily for 12 weeks
  Interventions: Drug: Placebo Control

INTERVENTIONS:
Drug: ADPS topical product — topical product
  Other Names: Active
  Arms: ADPS topical product
Drug: Placebo Control — topical product
  Other Names: vehicle
  Arms: Placebo Control

SUMMARY:
Safety and efficacy study in patients with acne vulgaris

DETAILED DESCRIPTION:
randomized, double-blind, placebo controlled, parallel-group, multiple-center study to evaluate the efficacy and safety of ADPS in the treatment of acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or non pregnant female aged ≥ 9 years with a clinical diagnosis of acne vulgaris

Exclusion Criteria:

* Female Subjects who are pregnant, nursing or planning to become pregnant during study participation.

Min Age: 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2016-10-03 (Actual); Primary Completion 2017-01-24 (Actual); Study Completion 2017-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catawba Research, Study Chair — http://catawbaresearch.com/contact/

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ADPS Topical Product | Placebo Control
Started | 147 | 147
Completed | 137 | 136
Not Completed | 10 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ADPS Topical Product | Placebo Control | Total
Number analyzed (Participants) | 147 | 147 | 294
Age, Categorical [Count of Participants; unit: Participants] — Population: The analysis population used for demographics excluded some subjects in baseline/randomized population.
  Participants
    number analyzed (Participants) | 146 | 141 | 287
    <=18 years | 57 | 58 | 115
    Between 18 and 65 years | 89 | 83 | 172
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.1 (8.29) | 22.4 (8.7) | 22.2 (8.48)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The analysis population used for demographics excluded some subjects in baseline/randomized population.
  Participants
    number analyzed (Participants) | 146 | 141 | 287
    Female | 83 | 98 | 181
    Male | 63 | 43 | 106
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The analysis population used for demographics excluded some subjects in baseline/randomized population.
  Participants
    number analyzed (Participants) | 146 | 141 | 287
    Hispanic or Latino | 75 | 69 | 144
    Not Hispanic or Latino | 71 | 72 | 143
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The analysis population used for demographics excluded some subjects in baseline/randomized population.
  Participants
    number analyzed (Participants) | 146 | 141 | 287
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 4 | 2 | 6
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 40 | 41 | 81
    White | 101 | 93 | 194
    More than one race | 1 | 5 | 6
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 147 | 147 | 294
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: The analysis population used for demographics excluded some subjects in baseline/randomized population.
  kg/m^2
    number analyzed (Participants) | 146 | 141 | 287
    (all) | 25.210 (6.6911) | 26.157 (6.8472) | 25.676 (6.7730)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline to Week 12 in the Inflammatory (Papules and Pustules) Lesion Counts on the Face
Time Frame: Baseline to week 12 (study day 84)
Population: The analysis population for efficacy excluded some subjects in baseline/randomized population.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage change in lesion counts
Arm/Group | ADPS Topical Product | Placebo Control
Number analyzed (Participants) | 146 | 141
percentage change in lesion counts | -60.84 [-64.31 to -57.36] | -62.17 [-65.71 to -58.62]
Statistical Analysis 1: Comparison: ADPS Topical Product vs Placebo Control; Test type: Superiority; p = 0.5947, ANOVA; LS Mean Difference = 1.33

2. Primary Outcome: Percent Change From Baseline to Week 12 in the Non-inflammatory (Open and Closed Comedones) Lesion Counts on the Face
Time Frame: Baseline to week 12 (study day 84)
Population: The analysis population for efficacy excluded some subjects in baseline/randomized population.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage change in lesion counts
Arm/Group | ADPS Topical Product | Placebo Control
Number analyzed (Participants) | 146 | 141
percentage change in lesion counts | -49.91 [-53.53 to -46.30] | -52.67 [-56.35 to -48.98]
Statistical Analysis 1: Comparison: ADPS Topical Product vs Placebo Control; Test type: Superiority; p = 0.2912, ANOVA; LS Mean Difference = 2.75

3. Primary Outcome: The Percentage of Subjects With a Clinical Response (IGA) of "Success" at Week 12 on the Face.
Description: Success was defined as an IGA score that was at least two grades less than the baseline assessment.
Time Frame: Baseline to Week 12 (study day 84)
Population: The analysis population for efficacy excluded some subjects in baseline/randomized population.
Measure: Number; unit: Percentage of subjects
Arm/Group | ADPS Topical Product | Placebo Control
Number analyzed (Participants) | 146 | 141
Percentage of subjects | 13.0 | 10.6
Statistical Analysis 1: Comparison: ADPS Topical Product vs Placebo Control; Test type: Superiority; p = 0.6920, Cochran-Mantel-Haenszel; Percent difference = 2.4

ADVERSE EVENTS:
Time Frame: 1 year
Description: An adverse event was defined as "Any untoward medical occurrence in a Subject or clinical-trial Subject administered a medicinal product and which does not necessarily have to have a causal relationship with this treatment", not any untoward or unfavorable medical occurrence in a participant " temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research" as defined by clinicaltrials.gov.
Arm/Group | ADPS Topical Product | Placebo Control
All-Cause Mortality (participants affected / at risk) | 0/146 | 0/141
Serious Adverse Events (participants affected / at risk) | 0/146 | 1/141
Other Adverse Events (participants affected / at risk) | 2/146 | 3/141
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ADPS Topical Product (N=146) | Placebo Control (N=141)
Spontaneous abortion (Product Issues) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ADPS Topical Product (N=146) | Placebo Control (N=141)
Nasopharyngitis (Infections and infestations) | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-02): https://cdn.clinicaltrials.gov/large-docs/36/NCT02935036/Prot_SAP_000.pdf